CLINICAL TRIAL: NCT02258217
Title: Tolerability of Acthar for the Treatment of Multiple Sclerosis Relapses (TAMS)
Brief Title: Tolerability of Acthar for the Treatment of Multiple Sclerosis in Relapses (TAMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014H0156
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2019-05

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Acthar 80 units subcutaneously for five consecutive days.
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — Is indicated for the treatment of acute exacerbations of multiple sclerosis in adults.
  Other Names: repository corticotropin

SUMMARY:
Tolerability of Acthar for the Treatment of Multiple Sclerosis Relapses (TAMS)

DETAILED DESCRIPTION:
We propose to conduct a prospective, single-center, open-label, single-arm study comparing tolerability of Acthar versus oral prednisone in the treatment of MS relapses. Potential subjects will be identified during routine clinical evaluations. If patient is determined to be having a study-defined MS relapse, they will be invited to participate in this study. After consent is obtained, the patient will complete the first page of the ARMS survey. If prior steroid use was deemed tolerable then only the first page of the ARMS will be collected and analyzed and these patients will complete their participation in the trial. Their data from the ARMS will provide an estimate as to the number of patients who self-report tolerability and efficacy issues with steroids. However, if patients self-report prior steroid intolerability, then they will advance into the Acthar treatment arm of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have volunteered and consented to participate in the study.
2. Subjects who have no contraindication to taking high dose, oral prednisone or Acthar.
3. Male or Female subjects age 18 or greater years of age.
4. Subjects with Relapsing Remitting Multiple Sclerosis (RRMS) based on 2010 McDonald Criteria.
5. Subjects without an active infection (Note: If a patient is found to have an uncomplicated UTI and agrees to start on appropriate antibiotic treatment, they can continue in the study).
6. Subjects who are experiencing a protocol defined MS relapse within two weeks of relapse onset.
7. Subjects who are able and willing to sign a consent form.

Exclusion Criteria:

1. Subjects who are less than 18 years of age.
2. Subjects with any contraindication to taking Acthar.
3. Subjects with an active infection other than an uncomplicated urinary tract infection (UTI) (subjects determined to have a UTI who agree to be treated with appropriate antibiotics will not be excluded).
4. Subjects with an immune deficiency.
5. Subjects with a history of any of the following conditions: gastrointestinal ulcers, diabetes mellitus, gestational diabetes, malignant hypertension or steroid induced psychosis.
6. Subjects who are pregnant or breastfeeding.
7. Subjects who are unable or unwilling to sign consent form.
8. Patient is unable or unwilling to participate in phone and clinic follow up.
9. Other factors that in the opinion of the Principal Investigator would exclude the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06-24 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron L Boster, MD, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth, Columbus, Ohio, United States

REFERENCES:
- [Background] Fox RJ, Bethoux F, Goldman MD, Cohen JA. Multiple sclerosis: advances in understanding, diagnosing, and treating the underlying disease. Cleve Clin J Med. 2006 Jan;73(1):91-102. doi: 10.3949/ccjm.73.1.91. PMID 16444920
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061
- [Background] Noseworthy JH, Lucchinetti C, Rodriguez M, Weinshenker BG. Multiple sclerosis. N Engl J Med. 2000 Sep 28;343(13):938-52. doi: 10.1056/NEJM200009283431307. No abstract available. PMID 11006371
- [Background] O'Brien JA, Ward AJ, Patrick AR, Caro J. Cost of managing an episode of relapse in multiple sclerosis in the United States. BMC Health Serv Res. 2003 Sep 2;3(1):17. doi: 10.1186/1472-6963-3-17. PMID 12952552
- [Background] Barnes D, Hughes RA, Morris RW, Wade-Jones O, Brown P, Britton T, Francis DA, Perkin GD, Rudge P, Swash M, Katifi H, Farmer S, Frankel J. Randomised trial of oral and intravenous methylprednisolone in acute relapses of multiple sclerosis. Lancet. 1997 Mar 29;349(9056):902-6. doi: 10.1016/s0140-6736(96)06453-7. PMID 9093250
- [Background] Morrow SA, Stoian CA, Dmitrovic J, Chan SC, Metz LM. The bioavailability of IV methylprednisolone and oral prednisone in multiple sclerosis. Neurology. 2004 Sep 28;63(6):1079-80. doi: 10.1212/01.wnl.0000138572.82125.f5. PMID 15452302
- [Background] La Mantia L, Eoli M, Milanese C, Salmaggi A, Dufour A, Torri V. Double-blind trial of dexamethasone versus methylprednisolone in multiple sclerosis acute relapses. Eur Neurol. 1994;34(4):199-203. doi: 10.1159/000117038. PMID 7915989
- [Background] Burton JM, O'Connor PW, Hohol M, Beyene J. Oral versus intravenous steroids for treatment of relapses in multiple sclerosis. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD006921. doi: 10.1002/14651858.CD006921.pub3. PMID 23235634
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Hobart J, Lamping D, Fitzpatrick R, Riazi A, Thompson A. The Multiple Sclerosis Impact Scale (MSIS-29): a new patient-based outcome measure. Brain. 2001 May;124(Pt 5):962-73. doi: 10.1093/brain/124.5.962. PMID 11335698
- [Background] Perrin Ross A, Williamson A, Smrtka J, Flemming Tracy T, Saunders C, Easterling C, Niewoehner J, Mutschler N. Assessing relapse in multiple sclerosis questionnaire: results of a pilot study. Mult Scler Int. 2013;2013:470476. doi: 10.1155/2013/470476. Epub 2013 May 26. PMID 23766909

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: ARMS (Assessing Relapses in Multiple Sclerosis) ADL Scores (Activities of Daily Living)
Description: Patient history of prior corticosteroid tolerability for the treatment of MS relapses. This will be determined based on patient completion of the ARMS survey at the baseline visit. Also, history of patients from the survey after treatment for the new relapse will be collected.
  The ARMS questionnaire (assessing relapses in multiple sclerosis) was developed by a panel of expert MS nurses. Part one consists of 7 questions designed to assess relapse symptoms, impact on activities of daily living, and response to past treatment for MS relapses. Part two consists of 7 questions to evaluate treatment response in terms of relief from symptoms, functioning and tolerability.
  ADL scores were calculated from Part 1 (new relapse), question 3 and Part 2 (after treatment of relapse), question 5 both specifically refer to ADL;
  Scale: ADL (Activities of Daily Living) Minimum value: 0 Maximum value: 9 Higher scores indicated better functioning/ improvement.
Time Frame: baseline visit & follow-up after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 30
score on a scale
  ADL (new relapse) | 3.1 (2.2)
  ADL (after treatment of relapse) | 4.9 (2.8)
Statistical Analysis 1: Comparison: Single Arm; We compared the two ADL scores measured in the same arm at different timepoints (new & after treatment). Null Hypothesis = Difference in means is = 0 Alternate Hypothesis = Difference in means is not = 0 We used the Paired t-test to compare the pre - post ADL scores; Test type: Equivalence — We created a difference in ADL score variable. This was calculated as follows: ADL score (new relapse) - ADL score (after treatment of current relapse) This difference score was tested for equivalence to 0 or not; p = 0.003, Paired t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-2.9 to -0.66], Standard Deviation 3.03

2. Primary Outcome: ARMS (Assessing Relapses in Multiple Sclerosis) RSH Scores (Return to Previous Health)
Description: Patient history of prior corticosteroid tolerability for the treatment of MS relapses. This will be determined based on patient completion of the ARMS survey at the baseline visit. Also, patients completed the survey after treatment for the new relapse. The ARMS questionnaire (assessing relapses in multiple sclerosis) was developed by a panel of expert MS nurses. Part one consists of 7 questions designed to assess relapse symptoms, impact on activities of daily living, and response to past treatment for MS relapses. Part two consists of 7 questions to evaluate treatment response in terms of relief from symptoms, functioning and tolerability.
  Part 1 (new relapse) & Part 2 (after treatment of new relapse), question 6 were used to calculate RSH;
  Scale: RSH (Return to previous health) Minimum value: -1 Maximum value: 10 Higher scores indicating a more complete return to previous state of health.
Time Frame: baseline visit & follow-up after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 27
score on a scale
  RSH (new relapse) | 4.6 (2.9)
  RSH (after treatment of new relapse) | 4.4 (3.2)
Statistical Analysis 1: Comparison: Single Arm; We compared the two RSH scores measured in the same arm at different time points (new & after treatment). Null Hypothesis = Difference in means is = 0 Alternate Hypothesis = Difference in means is not = 0 We used the Paired t-test to compare the pre - post RSH scores; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.99, Paired t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-1.22 to 1.22], Standard Deviation 3.09

3. Primary Outcome: ARMS (Assessing Relapses in Multiple Sclerosis) TCS Scores (Total Composite Scores)
Description: Patients completed the ARMS survey after treatment for the new relapse.The ARMS questionnaire (assessing relapses in multiple sclerosis) was developed by a panel of expert MS nurses. Part one consists of 7 questions designed to assess relapse symptoms, impact on activities of daily living, and response to past treatment for MS relapses. Part two consists of 7 questions to evaluate treatment response in terms of relief from symptoms, functioning and tolerability.
  The TCS score was calculated only for the time point after treatment of relapse. It was a sum of questions 4 (symptom improvement), 5 (ADL), and 6 (return to previous state of health (RSH)) were evaluated. Scores range from 0 to 30 units, with higher scores representing greater improvement/better functioning.
Time Frame: Follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 29
score on a scale | 14.3 (8.5)

4. Primary Outcome: ARMS (Assessing Relapses in Multiple Sclerosis) PCS Scores (Partial Composite Scores)
Description: Patient history of prior corticosteroid tolerability for the treatment of MS relapses. This will be determined based on patient completion of the ARMS survey at the baseline visit. Also, patients completed the survey after treatment for the new relapse.
  The ARMS questionnaire (assessing relapses in multiple sclerosis) was developed by a panel of expert MS nurses. Part one consists of 7 questions designed to assess relapse symptoms, impact on activities of daily living, and response to past treatment for MS relapses. Part two consists of 7 questions to evaluate treatment response in terms of relief from symptoms, functioning and tolerability.
  PCS was computed based on the sum of the ADL and RSH questions. The PCS was computed separately for Part 1 (new relapse) and Part 2 (after relapse treatment) and summarized descriptively; Higher scores indicating better functioning/greater improvement. The PCS scores were on a scale of 0 to 20 units.
Time Frame: baseline visit & follow-up after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 27
score on a scale
  PCS (New relapse) | 7.7 (3.3)
  PCS (after treatment of relapse) | 9.2 (5.6)
Statistical Analysis 1: Comparison: Single Arm; We compared the two PCS scores measured in the same arm at different timepoints (new & after treatment). Null Hypothesis = Difference in means is = 0 Alternate Hypothesis = Difference in means is not = 0 We used the Paired t-test to compare the pre - post PCS scores; Test type: Equivalence — We created a difference in PCS score variable. This was calculated as follows: PCS score (new relapse) - PCS score (after treatment of current relapse). This difference score was tested for equivalence to 0 or not; p = 0.03, Paired t-test, two sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.67 to -0.18], Standard Deviation 4.42

5. Primary Outcome: MSIS (Multiple Sclerosis Impact Scale) -29 Physical Score
Description: The MSIS-29 is a self-reported questionnaire in which MS patients answer a series of 29 questions designed to capture the impact of multiple sclerosis on their life over the past 2 weeks (11). Twenty of the 29 questions assess the physical impact of MS.
  The physical impact of MS was compared between pre and post phase using paired t-tests. Each question is answered with points ranging from 1 to 5. Higher score indicates worse outcome. The total MSIS physical score ranges from 20 to 100 points with lower points indicating better impact.
Time Frame: baseline visit & follow-up after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 30
score on a scale
  MSIS physical (new relapse) | 58.5 [23 to 90]
  MSIS physical (after treatment of new relapse) | 56 [20 to 91]
Statistical Analysis 1: Comparison: Single Arm; We compared the two MSIS physical scores measured in the same arm at different timepoints (new relapse & after treatment of relapse). Null Hypothesis = Difference in medians is = 0 Alternate Hypothesis = Difference in medians is not = 0 We used the Wilcoxon Signed rank test to compare the pre - post MSIS physical scores; Test type: Equivalence — We created a difference in MSIS physical score variable. This was calculated as follows: MSIS physical score (new relapse) - MSIS physical score (after treatment of current relapse) This difference score was tested for equivalence to 0 or not; p = 0.19, Wilcoxon Signed Rank test; Median Difference (Final Values) = 2.5

6. Primary Outcome: MSIS (Multiple Sclerosis Impact Scale) - 29 Psychological Score.
Description: The MSIS-29 is a self-reported questionnaire in which MS patients answer a series of 29 questions designed to capture the impact of multiple sclerosis on their life over the past 2 weeks (11). Twenty of the 29 questions assess the physical impact of MS and 9 questions assess the psychological impact of MS.
  The psychological impact of MS was compared between pre and post phase using paired t-tests.
  The psychological impact of MS was compared between pre and post phase using paired t-tests.
  The score was on a scale of 9 to 45 points for MSIS psychological score.
  Higher score indicate worse outcome.
Time Frame: baseline visit & follow-up after treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 30
score on a scale
  MSIS psychological(new relapse) | 29.4 [12 to 45]
  MSIS psychological(after treatment of new relapse) | 26.3 [9 to 45]
Statistical Analysis 1: Comparison: Single Arm; We compared the two MSIS psychological scores measured in the same arm at different timepoints (new relapse & after treatment of relapse). Null Hypothesis = Difference in means is = 0 Alternate Hypothesis = Difference in means is not = 0 We used the Paired t-test to compare the pre - post MSIS psychological scores; Test type: Equivalence — We created a difference in MSIS psychological score variable. This was calculated as follows: MSIS psychological score (new relapse) - MSIS psychological score (after treatment of current relapse) This difference score was tested for equivalence to 0 or not; p = 0.01, Paired t-test, 2 sided; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [0.74 to 5.45], Standard Deviation 6.3

7. Primary Outcome: EDSS (Expanded Disability Status Scale) Scores.
Description: This scaling score is obtained by performing a neurologic exam with specific attention to eight different neurologic functional systems: visual, pyramidal, cerebellar, bowel and bladder, cerebral, brainstem, sensory and other (10). The score is rated from zero (normal neurologic examination) to ten (death due to MS). This is the standard neurologic disability scale used in clinical trials for the evaluation of disability in patients with MS.
  These scores were compared between pre and post phase using paired t-tests.
Time Frame: baseline and at follow-up
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 13
score on a scale
  EDSS score (new relapse) | 3.5 [0 to 8]
  EDSS score (after treatment of new relapse) | 3.0 [0 to 7.5]
Statistical Analysis 1: Comparison: Single Arm; We compared the two EDSS scores measured in the same arm at different timepoints (new relapse & after treatment of relapse). Null Hypothesis = Difference in medians is = 0 Alternate Hypothesis = Difference in medians is not = 0 We used the Wilcoxon Signed rank test to compare the pre - post EDSS scores; Test type: Equivalence — We created a difference in EDSS score variable. This was calculated as follows: EDSS score (new relapse) - EDSS score (after treatment of current relapse) This difference score was tested for equivalence to 0 or not; p = 0.23, Wilcoxon Signed Rank test; Median Difference (Final Values) = 0 — The interquartile range for the median difference in EDSS scores is 0.0 to 0.5

8. Primary Outcome: SAGE (Self-administered Gerocognitive Exam) Scores
Description: The Self-Administered Gerocognitive Exam (SAGE) is designed to detect early signs of cognitive, memory or thinking impairments. It evaluates your thinking abilities and helps physicians to know how well your brain is working.
  It consists of 12 questions which are scored at different scales. The final SAGE score is calculated as a sum of these 12 questions and it ranges from 0 to 22.
  Higher score indicates better outcome.
Time Frame: baseline and follow-up
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 25
score on a scale
  SAGE (new relapse) | 21 [14 to 22]
  SAGE (after treatment of new relapse) | 21 [15 to 22]
Statistical Analysis 1: Comparison: Single Arm; We compared the two SAGE scores measured in the same arm at different time points (new relapse & after treatment of relapse). Null Hypothesis = Difference in medians is = 0 Alternate Hypothesis = Difference in medians is not = 0 We used the Wilcoxon Signed rank test to compare the pre - post SAGE scores; Test type: Equivalence — We created a difference in SAGE score variable. This was calculated as follows: SAGE score (new relapse) - SAGE score (after treatment of current relapse) This difference score was tested for equivalence to 0 or not; p = 0.44, Wilcoxon Signed Rank test; Median Difference (Final Values) = 0 — The interquartile range for the difference in medians is -1 to 0

9. Secondary Outcome: GASE Scale Questionnaire (Generic Assessment of Side Effects)
Description: Patients who reported a history of poor corticosteroid tolerability will be placed on Acthar and GASE scale will be given to assess tolerability to Acthar.
  We listed the number of times a symptom was reported and was attributable to the ACTHAR treatment
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 29
Participants
  Headache | 3
  Dry Mouth | 1
  Dizziness | 2
  Tachycardia, palpitation or arrhythmia | 1
  Breathing problems | 1
  Abdominal pain | 4
  Nausea | 4
  Diarrhea | 4
  Reduced Appetite | 1
  Increased appetite | 4
  Difficulties with urination | 2
  Skin rash or itching | 1
  Tendency to develop bruises | 1
  Sweating | 1
  Hot flashes | 1
  Fatigue, loss of energy | 2
  Insomnia, sleeping problems | 8
  Nightmares or abnormal dreams | 2
  Back pain | 1
  Agitation | 6
  Irritability | 6
  Depressed Mood | 3
  Anxiety, fearfulness | 1
  Further symptoms | 8

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No